CLINICAL TRIAL: NCT07135869
Title: Reliability and Discriminant Validity of a Mobile App for Detecting Muscle Fatigue in People With Cystic Fibrosis
Brief Title: Muscle Fatigue in People With Cystic Fibrosis: Insight From a Mobile App
Status: Recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Diego Ruiz-Cárdenas, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: CE042404
Record Dates: First submitted 2025-05-14; First posted 2025-08-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; Fatigue; Fatigability; Mobile app; Validity; Reliability; Muscle power; Strength; Peripheral muscle function
MeSH Terms: conditions — Cystic Fibrosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatigue protocol for cystic fibrosis: The one minute sit-to-stand test will be used as fatigue protocol.
  Interventions: Diagnostic Test: One minute sit-to-stand test
- Fatigue protocol for healthy controls: The one minute sit-to-stand test will be used as fatigue protocol
  Interventions: Diagnostic Test: One minute sit-to-stand test

INTERVENTIONS:
Diagnostic Test: One minute sit-to-stand test — The one minute sit-to-stand test will be used as acute fatigue protocol to generate fatigue.

SUMMARY:
Muscle fitness is an important component of health. For instance, the ability to resist to muscle fatigue development is important for daily functioning. Previous studies have suggested altered muscle function in people with cystic fibrosis. However, it is unclear whether such findings still apply in the modern era of CF. Several studies suggested that recent improvements in therapeutics, including CFTR modulators, may have positive effects on the skeletal muscles, potentially normalizing the ability to resist to muscle fatigue. However, no studies to date compared muscle fatigue between people with cystic fibrosis and healthy controls in a large sample of patients. One difficulty is that muscle fatigue assessment requires high-cost dynamometric instruments, which also leads to a gap between research and clinical practice. Our research group has created a mobile application based on video analysis of the chair rising test that reports values of time, velocity and power as reliable as devices found in a laboratory environment. The application has been shown to be valid and reproducible for measuring muscle fatigue in healthy people. However, a validation is necessary before recommending its use in people with cystic fibrosis.

DETAILED DESCRIPTION:
Objectives: To evaluate the reliability of a mobile app to detect muscle fatigability as decrease in performance after 1minSTS test in people with cystic fibrosis, and to analyze whether muscle fatigability is still increased in people with cystic fibrosis compared to healthy controls.

Methods: A discriminant validity and reliability study designed in accordance with the Guidelines for Reporting Reliability and Agreement Studies will be carried out. The study will include at least 34 participants diagnosed with cystic fibrosis and 34 healthy participants matched for age, sex, and physical activity level. A fatigue protocol will be carried out that will consist of chair rising as many times as possible for 60 seconds. A measurement will be carried out before (Pre), immediately after (Post) and one minute after (Post1min) the fatigue protocol through the mobile application (Sit to Stand App). The time, velocity and power values derived from the application will be used as fatigability indicators. The differences between the Pre and Post measurements will be indicative of performance fatigability, while the differences between the Post and Post1min measurements will be indicative of recovery. Heart rate will be recorded during the fatigue protocol and Post1min, as well as muscle and respiratory effort using the Borg CR10 scale. This experimentation will be repeated twice with a difference of 30 minutes in order to analyze the reliability of the measurements.

The sample size estimation was calculated using G*Power 3.1 software. An estimation was performed for each study objective, and the estimation requiring the largest sample size was selected for the study.

To analyze whether the level of muscle fatigability is reproducible, a minimum acceptable reliability of ρH0 ≥ 0.5 and an expected reliability of ρH1 ≥ 0.8 were selected. For a two-tailed test with a statistical power ≥ 80% and an alpha error of 0.05, the minimum required sample size was reported as 29 participants. To analyze whether mobile application detects muscle fatigability induced by the fatigue test, an expected moderate effect size (d ≥ 0.7) with a statistical power ≥ 80% and an alpha error of 0.05 was selected, resulting in a minimum desirable sample size of 34 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable.
* No changes in medication or pulmonary exacerbations within the two weeks prior to inclusion.
* Not requiring oxygen therapy during the test.
* No history of lung or liver transplants.

Exclusion Criteria:

* Any musculoskeletal conditions that could limit or influence test performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with cystic fibrosis, recruited from the registry of the Cystic Fibrosis Association of Murcia, and healthy control participants matched by age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rising Time | Twice separated by 30 minutes to assess reliability.
  Rising time derived from the mobile application (Sit to Stand App) will be carried out before (Pre), immediately after (Post) and one minute after (Post1min) the fatigue protocol. The differences between the Pre and Post measurements will be indicative of fatigability, while the differences between the Post and Post1min measurements will be indicative of recovery. We will follow the protocol published previously (https://doi.org/10.1007/s00421-024-05537-9).
Sit to Stand Velocity | Twice separated by 30 minutes to assess reliability.
  Velocity derived from the mobile application (Sit to Stand App) will be carried out before (Pre), immediately after (Post) and one minute after (Post1min) the fatigue protocol. The differences between the Pre and Post measurements will be indicative of fatigability, while the differences between the Post and Post1min measurements will be indicative of recovery. We will follow the protocol published previously (https://doi.org/10.1007/s00421-024-05537-9).
Sit to Stand Power | Twice separated by 30 minutes to assess reliability.
  Power derived from the mobile application (Sit to Stand App) will be carried out before (Pre), immediately after (Post) and one minute after (Post1min) the fatigue protocol. The differences between the Pre and Post measurements will be indicative of fatigability, while the differences between the Post and Post1min measurements will be indicative of recovery. We will follow the protocol published previously (https://doi.org/10.1007/s00421-024-05537-9).
One minute sit-to-stand test | Twice separated by 30 minutes to assess reliability.
  The one minute sit-to-stand test will be carried out according to the Guidance and standard operating procedures for functional exercise testing in cystic fibrosis (https://doi.org/10.1183/16000617.0029-2023). The number of repetitions performed during the test will be collected.

SECONDARY OUTCOMES:
Heart rate | Twice separated by 30 minutes to assess reliability.
  Heart rate will be recorded at rest, during the fatigue protocol, and after 1 minute of recovery.
Muscle effort | Twice separated by 30 minutes to assess reliability.
  Muscle effort will be recorded at rest, and after the fatigue protocol using the Borg CR10 scale.
Respiratory effort | Twice separated by 30 minutes to assess reliability.
  Respiratory effort will be recorded at rest, and after the fatigue protocol using the Borg CR10 scale.
Oxygen saturation | Twice separated by 30 minutes to assess reliability.
  Oxygen saturation (SpO2) will be recorded at rest, and after the fatigue protocol (Nadir SpO2).

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Ruiz-Cárdenas, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Asociación Murciana de Fibrosis Quistica, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saynor ZL, Gruet M, McNarry MA, Button B, Morrison L, Wagner M, Sawyer A, Hebestreit H, Radtke T, Urquhart DS; European Cystic Fibrosis Society Exercise Working Group. Guidance and standard operating procedures for functional exercise testing in cystic fibrosis. Eur Respir Rev. 2023 Aug 9;32(169):230029. doi: 10.1183/16000617.0029-2023. Print 2023 Sep 30. PMID 37558263
- [Background] Ruiz-Cardenas JD, Rodriguez-Juan JJ, Smart RR, Jakobi JM, Jones GR. Validity and reliability of an iPhone App to assess time, velocity and leg power during a sit-to-stand functional performance test. Gait Posture. 2018 Jan;59:261-266. doi: 10.1016/j.gaitpost.2017.10.029. Epub 2017 Oct 31. PMID 29102856
- [Background] Martinez-Garcia MDM, Rodriguez-Juan JJ, Ruiz-Cardenas JD. Influence of sex gap on muscle strength and functional mobility in patients with cystic fibrosis. Appl Physiol Nutr Metab. 2020 Apr;45(4):387-392. doi: 10.1139/apnm-2019-0484. Epub 2019 Sep 17. PMID 31526325
- [Background] Ruiz-Cardenas JD, Montemurro A, Del Mar Martinez-Garcia M, Rodriguez-Juan JJ. Concurrent and discriminant validity and reliability of an Android App to assess time, velocity and power during sit-to-stand test in community-dwelling older adults. Aging Clin Exp Res. 2023 Aug;35(8):1631-1640. doi: 10.1007/s40520-023-02451-6. Epub 2023 Jun 12. PMID 37306926
- [Background] Souron R, Ruiz-Cardenas JD, Gruet M. The 1-min sit-to-stand test induces a significant and reliable level of neuromuscular fatigability: insights from a mobile app analysis. Eur J Appl Physiol. 2024 Nov;124(11):3291-3301. doi: 10.1007/s00421-024-05537-9. Epub 2024 Jun 20. PMID 38900202
- [Background] Gruet M, Troosters T, Verges S. Peripheral muscle abnormalities in cystic fibrosis: Etiology, clinical implications and response to therapeutic interventions. J Cyst Fibros. 2017 Sep;16(5):538-552. doi: 10.1016/j.jcf.2017.02.007. Epub 2017 Mar 2. PMID 28262570